CLINICAL TRIAL: NCT01503190
Title: A Translational Study of the Interactions Between Prior Pregnancy and the Biologic Subtype of Breast Cancer in Defining the Cancer: Host Immunologic Interaction
Brief Title: The Immune System's Response to Young Women's Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0583.cc
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Cancer and Pregnancy
Keywords: Breast Cancer; Young Women; Pregnancy Associated Breast Cancer; Pregnancy; Premenopausal Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue, Blood and urine may be collected from subjects who were recently diagnosed. Subjects who were diagnosed after treatment begins or has ended will only be eligible for tissue donation section of study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study plans to learn more about the immune system's response to breast cancer in young women.

DETAILED DESCRIPTION:
The investigators will be looking at the level of immune suppression in different types of breast cancer. The investigators will use blood, urine, and tissue samples from patients with Pregnancy Associated Breast Cancer (PABC) versus non-PABC, as well as comparing different types of breast cancer. If tissue sampling permits, the investigators may use some of the breast cancer tissue to develop models for human cancer for drug targeting. Understanding the immune response and suppression in different types of cancer will help us understand mechanisms involved in breast cancer better and help the investigators in developing new treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Females >18.
2. Histological or cytological confirmation of breast cancer.
3. For patients diagnosed with needle core or excisional biopsy, formalin-fixed paraffin embedded tumor blocks or unstained slides should be available or planned to be available after upcoming procedure.
4. Patient should be willing to have fresh and/or fresh frozen tissue collected at time of core biopsy, definitive breast cancer surgery or clinically planned breast cancer metastasis biopsy/resection for research purposes as part of study procedures, if a procedure is in the future planning of the patient's treatment.
5. Any clinical stage allowed.
6. Written informed consent obtained prior to any initiation of study procedures in the case of subjects consented in clinic. Subjects consented outside of UCH, VVMC or SCC will be consented by phone and verbal informed consent will be obtained prior to any initiation of study procedures.
7. Women treated at UCH, VVMC or SCC may be pregnant. Other participants are excluded for safety reasons.
8. Women who have commenced or completed their breast cancer treatment may join this study by consenting to a retrospective tissue donation only consent of the protocol.
9. Women who receive their care at a facility other than UCH, VVMC or SCC may join this study. These women will be consented utilizing the phone consent and will receive a copy of the consent in the mail, or they will consent online and print a copy of their online consent.

Exclusion Criteria:

1. Known significant autoimmune condition [ie Lupus, Crohne's disease or Rhuematoid Arthritis], chronic oral steroid use, use of systemic immunomodulatory prescription drugs for any medical condition.
2. The presence of other comorbid conditions known to significantly impact immune function, (such as: type I diabetes, uncontrolled adult onset diabetes, severe COPD, uncontrolled infection or known HIV infection.)
3. Underlying psychiatric condition which would, in the opinion of the investigator, preclude compliance with study requirements
4. Subjects with a history of other malignancy besides current diagnosis of breast cancer who were diagnosed and treated within the last 5 years are excluded, with exception of cervical cancer definitively treated more than 2 years ago or non-melanomatous skin cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is restricted by gender due to the population of interest being women with pregnancy associated breast cancer and appropriately matched age controls.
Study Population: Women over the age of 18 who have been diagnosed with breast cancer. Women over age 46 will serve as controls. Need not be in active treatment.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2009-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Throughout study participation
  Prospective cohort study.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Borges, MD, MMSc, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - University of Colorado Denver, Aurora, Colorado
  - Denver Health Hospital Authority, Denver, Colorado
  - UCHealth Cherry Creek Medcial Center, Denver, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - UCHealth Lone Tree Medical Center, Lone Tree, Colorado

IPD SHARING:
Plan to Share IPD: No